CLINICAL TRIAL: NCT07230899
Title: A Cluster Randomized Controlled Trial of Cognitive Behavioural Therapy for Insomnia Among Young People With Moderate Level of Mental Distress in Hong Kong
Brief Title: Cognitive Behavioural Therapy for Insomnia Among Young People With Moderate Level of Mental Distress in Hong Kong
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); The Boys' and Girls' Clubs Association of Hong Kong (Other); Caritas Medical Centre, Hong Kong (Other); Hong Kong Christian Service (Other); Neighbourhood Advice-Action Council (Other); St. James' Settlement (Other); Tung Wah Group of Hospitals (Other); Hong Kong Young Women's Christian Association (Other); Yan Oi Tong (Unknown); The Salvation Army, Hong Kong and Macau Command (Other); Hong Kong Playground Association (HKPA) (Unknown); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Hong Kong Children and Youth Services (HKCYS) (Unknown); Hong Kong Federation of Youth's Group (HKFYG) (Other); Chinese YMCA of Hong Kong (Unknown)
Responsible Party: Principal Investigator, Dr. Christy Lai-ming Hui, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250818-002-000
Record Dates: First submitted 2025-08-27; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Mental Distress; Insomnia
Keywords: cluster randomized controlled trial; cognitive behavioural therapy for insomnia; youths; mental distress
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBTi Intervention (Active Comparator): The CBTi program, designed to improve youths' sleep quality, comprises six sessions scheduled to be delivered over a six-week period. The intervention will be conducted in a small-group format (4 or above participants per group). Each session is one hour long and is led by a trained LevelMind@JC worker. All sessions will be delivered in a face-to-face format by frontline social or youth workers who have undergone training by a clinical psychologist ensuring they possess the necessary expertise to effectively implement the CBTi intervention.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Waitlist Control (No Intervention): Participants allocated to the waitlist control group will wait for 10 weeks (6 + 4 weeks) before receiving the CBTi intervention

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Participants will receive the Cognitive Behavioral Therapy for Insomnia designed to improve youths' sleep quality.
  Arms: CBTi Intervention

SUMMARY:
This cluster randomized controlled trial (cRCT) aims to evaluate the effectiveness of a Cognitive Behavioral Therapy for Insomnia (CBTi) intervention in enhancing sleep quality, overall quality of life, functional ability, and reducing mental distress among at-risk youths in Hong Kong. Participants are youths with moderate mental health concerns, indicated by K6 scores ranging from 11 to 14.

The study involves seven clusters, each based on community hubs, which will be randomly assigned to either the intervention group or a wait-list control group. Clusters assigned to the intervention group will receive six weekly face-to-face sessions led by trained youth workers. Control clusters will receive the same intervention after the initial follow-up period.

Participants will be evaluated at baseline, post-intervention, and one-month follow-up. An interim analysis is built for the sake of evaluation of the collected data from the ongoing trial, in which the primary research question is addressed, and which has the potential for modifying the conduct of the study. Furthermore, a qualitative follow-up will be conducted after the trial, involving both participants and the workers delivering the CBTi intervention. This qualitative component aims to gather feedback on participants' experiences, and inform potential revisions to enhance future implementation.

It is hypothesized that youths receiving the CBTi intervention will show significantly greater improvements in sleep quality, quality of life, and functioning, along with reductions in mental distress, as well as depressive and anxiety symptoms, compared to those in the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* JC LevelMind @ Community users at risk for mental distress (Tier 2), with K6 scores ranging from 11 to 14
* Aged between 12 and 24 years
* Insomnia Severity Index (ISI) score greater than 7
* Sufficiently proficient in Chinese to comprehend verbal instructions
* Able to provide written informed consent (parental consent for participant aged 12-17)

Exclusion Criteria:

* Known diagnosis of intellectual disability
* Organic brain disorder
* Established psychiatric diagnosis
* Current substance abuse
* Receiving other structured psychological therapies such as module-based psychological therapy, mentalization-based therapy, low-intensity online interventions, cognitive-behavioral therapy, narrative therapy, mindfulness, or art-informed therapy within the hub setting or any others outside the hub setting
* Presence of current or active suicidal ideation or attempts

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 770 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality and Disturbance | Baseline, 6-week, 10-week
  Pittsburgh Sleep Quality Index Scale (scores range from 0 to 21 where a higher score indicate poorer sleep quality, and a score greater than 5 suggesting significant sleep difficulties)
Insomnia Severity | Baseline, 6-week, 10-week
  Insomnia Severity Index Scale (scores range from 0 to 28 where a higher score indicates greater insomnia severity and a score of 7 or less suggested no clinical insomnia)

SECONDARY OUTCOMES:
Psychological Distress | Baseline, 6-week, 10-week
  The 6-item Kessler Psychological Distress Scale (scores range from 0 to 24 where a higher score indicates a worse outcome)
Depression | Baseline, 6-week, 10-week
  The 9-item Patient Health Questionnaire (scores range of 0 to 27 where a higher score indicates a worse outcome)
Depression and Anxiety Symptoms | Baseline, 6-week, 10-week
  Depression Anxiety Stress Scales (scores range from 0 to 63 where a higher score indicates more severe symptoms)
Anxiety | Baseline, 6-week, 10-week
  The 7-item Generalized Anxiety Stress Scale (scores range from 0 to 21 where a higher score indicates a worse outcome)
Social and Occupational Functioning | Baseline, 6-week, 10-week
  Social and Occupational Functioning Assessment Scale (scores range from 0 to 100 where a higher score indicates a better outcome)
Health-related Quality of Life | Baseline, 6-week, 10-week
  The 12-item Short-Form 12 Health Survey (scores range from 0 to 100 where a higher score indicates a better outcome)
Health-related Quality of Life | Baseline, 6-week, 10-week
  The Short Form 6-Dimension (scores range from 0 to 1 where a higher score indicates a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Lai Ming Hui, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No